CLINICAL TRIAL: NCT06078774
Title: Redesigning Pediatric Primary Care Obesity Treatment: Virtual House Calls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20026673
Record Dates: First submitted 2023-08-28; First posted 2023-10-12 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Obesity, Pediatric
Keywords: Obesity; House Calls; Pediatric Primary Care; Virtual; Telehealth
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Health Coach - Parent/Child Dyad (Experimental): Focuses on providing personalized care conveyed in an integrated and visually demonstrated way for parent-child pairs. Healthy lifestyle changes and behaviors covered in sessions are designed to initiate and maintain behavior change in nutrition and physical activity with BMI improvement.
  Interventions: Behavioral: Virtual Health Coach

INTERVENTIONS:
Behavioral: Virtual Health Coach — Dyads first session will be 60-minutes, totaling 1 hour. Dyads will participate in weekly 30-minute sessions for weeks 2-12, totaling 5.5 hours.
  Dyads will participate bi-weekly 30-minute sessions for 12 weeks, totaling 3 hours.
  Dyads will participate in weekly 30-minute exercise sessions for 24-weeks, totaling 12 hours.
  Children will have 3, 30-minute visits with their primary care physician (PCP) every 3 months, totaling 1.5 hours.
  Parents will have three, 60-minute individual sessions, totaling 3 hours. Total study duration is 24 weeks, with a total of 26 contact hours.
  Sessions follow a behavior therapy approach, including guided goal-setting, self-monitoring, identifying barriers and solutions, contingency management, stimulus control, dealing with setbacks, maintenance and relapse prevention. Weight is assessed weekly by coaches, with MI-consistent, autonomy-supportive feedback provided. Parent sessions will focus on ways to support their child's weight management.

SUMMARY:
This study examines a redesign of pediatric primary care overweight/obesity treatment, augmenting typical in-person visits with: (1) direct-to-patient video telehealth to tailor counseling advice to families, (2) that leverages certified health coaches as a part of the care team, and (3) creates skills building in real-time within the home environment.

DETAILED DESCRIPTION:
Investigators will recruit children with an elevated body mass index (BMI) (85th to <99th percentile) and a parent. Dyads will participate in a 24-week intervention with a total of 26 contact hours. Dyads will participate in weekly education sessions for the first 12 weeks and bi-weekly sessions for the remaining 12 weeks. Additionally, dyads will participate in weekly exercise sessions.

Assessments will consist of anthropometric measures, psychological surveys, and nutritional evaluations. Assessments will be completed at baseline, 3-months and 6-months.

ELIGIBILITY:
Inclusion Criteria:

Children:

* Ages 9-13 years
* BMI 85th to <99th percentile
* Must be a patient within Health System Pediatric Primary Care
* Must be English or Spanish speaking

Parent:

-Must be English or Spanish speaking

Exclusion Criteria:

Children:

* Cannot have an emotional, social, or physical disability that would prevent them from participating in the protocol
* Non-English or Non-Spanish speaking
* Cannot have a medical condition resulting in unintentional weight gain (i.e. Prader Willi)
* Females cannot be pregnant
* In addition, children will potentially be excluded from participation if they have a positive screen during an interview led pre-screening eating disorder questionnaire

Parent:

-Non-English or Non-Spanish speaking

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Bean, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth Universiy, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the trial occurred from January 2024 through August 2024. Recruitment methods included physician referrals and direct patient messaging with the electronic health record.
Groups:
- Child: Children that participated in the Virtual Housecalls behavioral intervention with their parent.
- Parent: Parents that participated in the Virtual Housecalls behavioral intervention with their child.
Period: Overall Study
Arm/Group | Child | Parent
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Child | Parent | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (1.8) | 40.6 (5.8) | 26.4 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 1 | 2 | 3
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.99 (3.22) | 33.45 (3.83) | 29.72 (5.16)

OUTCOME MEASURES:

1. Primary Outcome: Recruitment of Participants.
Description: Percentage of participants recruited compared to goal sample size.
Time Frame: 6 months
Population: The Overall Number of Participants Analyzed reflects the target enrollment number and the data reported reflects the actual number of participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Child | Parent
Number analyzed (Participants) | 50 | 50
Participants | 5 | 5

2. Primary Outcome: Retention of Participants
Description: Ability to retain 70% of participants at primary end point.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Child | Parent
Number analyzed (Participants) | 5 | 5
Participants | 5 | 5

3. Primary Outcome: Number of Participants Who Reported Being Satisfied With the Intervention
Description: Measured in an exit interview. Participants were asked if they benefited from the program.
Time Frame: 6 months
Population: Only participants who participated in an exit interview were included in this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Child | Parent
Number analyzed (Participants) | 3 | 3
Participants | 3 | 3

4. Secondary Outcome: Body Mass Index Change
Description: Body Mass Index change (kg/m2) from baseline to 6-months for child and parent. National Health and Nutrition Examination Survey (NHANES) Anthropometry methods were used to measure height and weight to calculate Body Mass Index (BMI).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Child | Parent
Number analyzed (Participants) | 5 | 5
kg/m^2 | 1.07 (1.05) | -0.43 (1.18)

5. Secondary Outcome: Adolescent Reported Authoritative Parenting Style
Description: The Authoritative Parenting Index (API) was used to assess adolescent-report of authoritative parenting style. Scores range from 16-64 with higher scores indicating the adolescent perceives their parent to have a higher level of authoritative parenting behavior. Results reflect the adolescent's perception on their parent (mom or dad) who participated in the study.
Time Frame: Baseline, 3-, and 6-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Child
Number analyzed (Participants) | 5
units on a scale
  Baseline | 26.80 (6.54)
  3-months | 26.40 (2.41)
  6-months | 27.60 (4.93)

6. Secondary Outcome: Parent Reported Parenting Style
Description: The Parenting Styles and Dimension Questionnaire (PSDQ) was administered to parents to assess parent self-report of authoritative parenting style. Results reflect the participating parent's perception of their parenting style. Scores range from 1-5 with higher scoring indicating a greater frequency of authoritative parenting behaviors.
Time Frame: Baseline, 3-, and 6-months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Parent: Parents that participate in the Virtual Housecalls behavioral intervention with their child.
Arm/Group | Parent
Number analyzed (Participants) | 5
units on a scale
  Baseline | 4.16 (0.51)
  3-month | 4.2 (0.69)
  6-month | 4.25 (0.71)

7. Secondary Outcome: Dietary Intake
Description: Child participants completed a 24-hour food recall using the Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool. Total energy intake is reported from the 24-hour recall.
Time Frame: Baseline, 3-, and 6-months
Measure: Mean (Standard Deviation); unit: kilocalories
Arm/Group | Child
Number analyzed (Participants) | 5
kilocalories
  Baseline | 1606 (440)
  3-month | 1997 (1143)
  6-month | 1224 (385)

8. Secondary Outcome: Physical Activity.
Description: Engagement in physical activity self-reported by the Patient-Centered Assessment and Counseling for Exercise Plus Nutrition (PACE+) questionnaire. The measure is scored by averaging responses with a range of 0-7. Higher scores (5-7) indicate meeting activity guidelines.
Time Frame: Baseline, 3-, and 6-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Child
Number analyzed (Participants) | 5
units on a scale
  Baseline | 3.7 (1.6)
  3-month | 4.3 (1.6)
  6-month | 3.5 (1.3)

9. Secondary Outcome: Parent Reported Sleep Duration for Child
Description: Parents completed a subset of questions from the National Health and Nutrition Examination Survey (NHANES) regarding their child's sleep behaviors. Data is reported sleep duration (hours) for child on weekdays/school days.
Time Frame: Baseline, 3-month, and 6-month
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Child
Number analyzed (Participants) | 5
hours
  Baseline | 8.45 (1.12)
  3-month | 8.55 (1.303)
  6-month | 9.10 (0.96)

10. Secondary Outcome: Home Food Environment.
Description: The Home Food Inventory (HFI) was used to assess the availability of types of food in the home and calculate an overall obesogenic score. Scores range from 0-60, with high scores indicating a more obesogenic food environment.
Time Frame: Baseline, 3-, and 6-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent
Number analyzed (Participants) | 5
units on a scale
  Baseline | 15.40 (14.98)
  3-month | 10.60 (1.52)
  6-month | 11.20 (3.27)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Child | Parent
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT06078774/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT06078774/ICF_001.pdf